CLINICAL TRIAL: NCT03625726
Title: Ex Vivo Study of the Role of Soluble Endothelial Protein C Receptor in Cirrhosis-associated Hypercoagulability State
Brief Title: Rôle of the Soluble Endothelial Protein C Receptor in Cirrhosis-associated Hypercoagulability State (EXERCISE)
Acronym: EXERCISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: CHU-403; 2017-A00931-52 (Other: 2017-A00931-52)
Record Dates: First submitted 2018-07-30; First posted 2018-08-10 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Cirrhosis
Keywords: cirrhosis; hypercoagulability; thrombin generation assay; soluble Endothelial Protein C Receptor
MeSH Terms: conditions — Fibrosis; Thrombophilia | interventions — In Vitro Techniques

STUDY DESIGN:
Intervention Model Description: Exploratory, cross-sectional, case-control pathophysiology study, based on ex vivo treatment of blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with cirrhosis (Experimental): pathophysiology study, blood sample
  Interventions: Biological: Thrombin generation assay (in vitro)
- healthy volunteers (Placebo Comparator): pathophysiology study, blood sample
  Interventions: Biological: Thrombin generation assay (in vitro)
- patients with hepatocellular carcinoma (Placebo Comparator): pathophysiology study, blood sample
  Interventions: Biological: Thrombin generation assay (in vitro)

INTERVENTIONS:
Biological: Thrombin generation assay (in vitro) — One blood sample.

SUMMARY:
Cirrhosis is a condition in which the liver does not function properly due to long-term damage. This damage is characterized by the replacement of normal liver tissue by scar tissue.

The liver carries out several necessary functions, including synthesis of proteins participating in blood coagulation process. Some of these proteins contribute to coagulation and others make blood more fluid. In healthy people there is a balance between the two.

In cirrhotic patient, there is an imbalance inducing hypercoagulation (hypercoagulability state). Cirrhotic patients are so known to be at risk of vein thrombosis (for example portal vein thrombosis: clot in hepatic vein).

Mechanisms leading to this imbalance are unclear. Studies need to be completed to improve patient's management.

The EPCRs (Endothelial Protein C Receptor soluble) takes part in blood coagulation process. Previous studies have shown that blood levels of EPCRs are increased in patients with cirrhosis.

The primary purpose of the study is to evaluate if the EPCRs could play a role in cirrhosis-associated hypercoagulability state.

DETAILED DESCRIPTION:
Three groups will be constitued: one with cirrhotic patients, one with healthy volunteers, and one with patients with hepatocellular carcinoma, a form of liver cancer (previous studies have also shown that blood levels of EPCRs are increased in these patients).

All participants will undergo a unique visit at hospital. An informed consent will be obtained before any related study procedures*.

* procedures: physical examination (including height, weight, waist measurement), vital signs (blood pressure, heart rate, temperature), medical history, concomitant medication, blood sample.

ELIGIBILITY:
Patients with cirrhosis

Inclusion criteria :

* Male, age 18 or older
* Cirrhosis, defined by: prothombin time ≤ 70% +/- liver dysmorphism +/- Fibroscan > 12.5 kPa +/- histology +/- portal hypertension associated with hepatocellular insufficiency
* Cirrhosis associated with hepatitis B or C, or alcoholic liver disease, or non alcoholic steato hepatitis
* Measurable portal flow by ultrasound doppler
* Child Pugh score A,B or C, without acute infection or acute bleeding
* Signed written informed consent
* Affiliation to french social security system

Exclusion criteria :

* Known history of vein thrombosis
* Known family history (in first-degree relative) of spontaneous thrombosis
* Partial or complete portal system vein thrombosis
* Uncontrolled infection after 7-day course of antibiotics
* Anticoagulant intake
* Hepatocellular carcinoma
* Protected or deprived of liberty adult
* Any medical or surgical history that could interfere with the study, as judged by the investigator
* Blood transfusion within 7 days
* Participation in a clinical trial for drug

Healthy volunteers

Inclusion criteria :

* Male, age 18 or older
* Body Mass Index between 18 and 30 kg/m2
* Normal physical examination
* Willing and able to comply with requirements of the study
* Agree to be registered in the french national registry for healthy volunteers
* Signed written informed consent
* Affiliation to french social security system

Exclusion criteria :

* Any medical or surgical history that could interfere with the study, as judged by the investigator
* Participation in a clinical trial for drug
* Protected or deprived of liberty adult
* Known history of vein thrombosis
* Known family history (in first-degree relative) of spontaneous thrombosis
* Anticoagulant intake

Patients with hepatocellular carcinoma (HCC)

Inclusion criteria :

* Male, age 18 or older
* Histological diagnosis of HCC, or use of BCLC criteria for diagnosis
* Treatment naïve HCC
* Measurable portal flow by ultrasound doppler
* For patients with cirrhosis: Child Pugh score A,B or C, without acute infection or acute bleeding
* Signed written informed consent
* Affiliation to french social security system

Exclusion criteria :

* Known history of vein thrombosis
* Known family history (in first-degree relative) of spontaneous thrombosis
* Partial or complete portal system vein thrombosis
* For patients with cirrhosis: uncontrolled infection after 7-day course of antibiotics
* Anticoagulant intake
* Protected or deprived of liberty adult
* Any medical or surgical history that could interfere with the study, as judged by the investigator
* Blood transfusion within 7 days
* Prior treated malignancy within the previous 2 years (except basal cell and squamous cell skin cancer, and superficial bladder cancer)
* Participation in a clinical trial for drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Thrombin generation assay (area under the curve/ Endogenous Thrombin Potential) with thrombomodulin. | 24 months

SECONDARY OUTCOMES:
Thrombin generation assay parameters : peak height | 24 months
Thrombin generation assay parameters : lag time | 24 months
Thrombin generation assay parameters : time to peak | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Armand ABERGEL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France